CLINICAL TRIAL: NCT01464606
Title: International Pleuropulmonary Blastoma (PPB) Treatment and Biology Registry Protocol
Brief Title: International Pleuropulmonary Blastoma (PPB) Treatment and Biology Registry
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Principal Investigator, Kris Ann Schultz, M.D., Children's Hospitals and Clinics of Minnesota
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PPB Reg Tx-Biol-001
Record Dates: First submitted 2011-09-29; First posted 2011-11-03 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pleuropulmonary Blastoma
Keywords: pleuropulmonary blastoma; pediatric; lung cysts
MeSH Terms: conditions — Pleuropulmonary blastoma; Cystic Disease Of Lung | interventions — Vincristine; Dactinomycin; Cyclophosphamide; Ifosfamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Type I PPB therapy (Experimental): PPB Type I therapy: All patients will be treated with surgery. Chemotherapy after surgery is per the treating physician(s) discretion. If chemotherapy is used the Registry will suggest that it be combination chemotherapy with Vincristine, Dactinomycin, Cyclophosphamide (VAC).
  Interventions: Drug: Vincristine; Drug: Dactinomycin; Drug: Cyclophosphamide
- Types II and III PPB therapy (Experimental): Combination chemotherapy with Ifosfamide, Vincristine, Dactinomycin and Doxorubicin ("IVADo"). Second look and possible 3rd look surgery may be required. Radiation therapy is recommended only for residual disease after maximum surgery.
  Interventions: Drug: Vincristine; Drug: Dactinomycin; Drug: Cyclophosphamide; Drug: Ifosfamide; Drug: Doxorubicin

INTERVENTIONS:
Drug: Vincristine — ≥ 3 years: 1.5 mg/m2 IV x 1 (maximum dose 2 mg)
  Other Names: Vincristine; Oncovin
Drug: Dactinomycin — ≥ 3 years: 0.045 mg/kg (maximum dose 2.5 mg) IV X 1
  Other Names: Actinomycin-D
Drug: Cyclophosphamide — ≥ 3 year: 1.2 gm/m2/dose IV as 1 hr infusion with IV fluids
  Other Names: Cytoxan
Drug: Ifosfamide — ≥ 3 years: 3 g/m2/dose IV over 3 hours on Days 1, 2, (6 g/m2/cycle)
  Other Names: Ifos
  Arms: Types II and III PPB therapy
Drug: Doxorubicin — ≥ 3 years: 30 mg/m2/dose IV over 30 min, Days 1, 2 (60 mg/m2/cycle)
  Other Names: Adriamycin
  Arms: Types II and III PPB therapy

SUMMARY:
Pleuropulmonary Blastoma (PPB) is very rare and there is no established "standard" or "best" therapy. For many years, children with PPB around the world have been treated according to decisions made case-by-case in many different hospitals by many different physicians. No treatment has been tested in a large group of PPB patients.

The goal is to treat many children with one treatment program and to learn the results of the treatment.

DETAILED DESCRIPTION:
This Registry will collect family medical history and establishes a collection of specimens from PPB patients and their parents for future research. Primary goals of the biology research are (1) to identify new scientific ways to learn about PPB and the best way to treat it in the future and (2) to establish a collection of PPB biologic specimens for future research.

Background: PPB is a rare cancer of the lung presenting in early childhood, mostly from birth to age ~72 months. PPB occurs within the lung or between the lung and the chest wall. There are three forms of PPB called Types I, II, and III PPB. Children with Type I PPB require surgery and sometimes chemotherapy. Children with Types II and III PPB, require surgery, chemotherapy and sometimes radiation therapy. Because there has never been a consensus as to the best treatment for PPB, the Registry will provide treatment guidelines. It is the goal of the Treatment and Biology Registry that by offering specific regimens the Registry will be able to prospectively review and analyze the regimen for the first time.

Design:

* Diagnostic central pathology review will be required for patients who will be prospectively evaluated.
* This Treatment Registry will offer surgery and chemotherapy regimen guidelines, and optional radiation therapy guidelines for prospectively enrolled patients.
* The Treatment and Biology Registry will create a PPB biologic specimens reference bank for tumor.

Methods:

* For Type I PPB, surgery is necessary. Some doctors use chemotherapy after surgery. If chemotherapy is used the Registry will suggest that it be combination chemotherapy with vincristine, dactinomycin, cyclophosphamide (VAC ).
* For Types II and III PPB patients surgery is necessary, followed by chemotherapy. The Registry will suggest that subjects receive combination chemotherapy with Ifosphamide, Vincristine, Actinomycin-D and Doxorubicin (IVADo). Second look and possible 3rd look surgery may be required. Radiation therapy is recommended only for residual disease after maximum surgery.

Analysis: Statistical data analysis will include only centrally confirmed cases. Additionally only patients with PPB Type II or Type III who were enrolled and treated with IVADo as per the regimen will be compared to historical controls. No statistical analysis is planned for patients with Type I PPB. Future treatment will be compared to the IVADo regimen in order to measure improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Age : Patients from birth to < 21 years of age at the time of diagnosis will be included in the Treatment and Biology Registry.

   Patients of any age will be included in the Associated Diseases arm of this study.
2. Pathology Diagnosis: Patients with newly-diagnosed PPB Types I, II or III. Diagnosis is made by the local pathologist. Real-time central pathology review is encouraged but is not required. All cases must be submitted for central pathology review. Only centrally-reviewed cases confirmed as PPB will be analyzed prospectively.

   Cases in which the initial diagnosis is "suggestive" or "supportive" of PPB, but not diagnostic, and in which later resection specimens, including resections following chemotherapy, confirm a PPB diagnosis will be included. Patients diagnosed by fine needle aspiration biopsy will be included only if a later resection specimen, including resections following chemotherapy, is diagnostic of PPB.

   Diagnostic pathology for cases of diseases associated with PPB will also require registry central pathology review.
3. Prior Therapy: PPB Type I: All patients are eligible and will be followed in the study.

   PPB Types II or III: Newly-diagnosed Types II and III PPB patients will be included in the Treatment and Biology Registry.

   DICER1-related condition and DICER1 gene mutation: all patients are eligible and will be followed in the study.
4. Prior corticosteroid therapy is allowed.
5. Patients who have received other chemotherapy regimens or radiation therapy will not be statistical analysis.
6. Types II and III PPB patients with PRIOR Type I PPB diagnosis: Types II and III PPB cases which are recurrences of an earlier Type I PPB are included.
7. Informed consent by patient or parent/guardian. (also, where appropriate: assent and HIPPA consent)

Exclusion Criteria:

1. Inability of patient, or parent/guardian to obtain informed consent.
2. Patients who have their PPB diagnosed ruled out by Registry central pathology review.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2009-12-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 5 years
  The primary endpoint for statistical analysis will be time from start treatment to an event, defined as the occurrence of progression or recurrence of PPB, occurrence of a second malignant neoplasm, or death from any cause that is at least possibly related to the original disease or treatment.

SECONDARY OUTCOMES:
Overall response to chemotherapy, and survival | 5 years
  Secondary endpoints will the best overall response to chemotherapy among patients with radiographically measurable tumor following initial surgery or biopsy, and time to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Kris Ann P Schultz, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Anne K Harris, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Hill DA, Ivanovich J, Priest JR, Gurnett CA, Dehner LP, Desruisseau D, Jarzembowski JA, Wikenheiser-Brokamp KA, Suarez BK, Whelan AJ, Williams G, Bracamontes D, Messinger Y, Goodfellow PJ. DICER1 mutations in familial pleuropulmonary blastoma. Science. 2009 Aug 21;325(5943):965. doi: 10.1126/science.1174334. Epub 2009 Jun 25. PMID 19556464
- See also: Pleuropulmonary Blastoma Registry web site — http://www.ppbregistry.org